CLINICAL TRIAL: NCT02442297
Title: Phase I Study of Intracranial Injection of T Cells Expressing HER2-specific Chimeric Antigen Receptors (CAR) in Subjects With HER2-Positive Tumors of the Central Nervous System (iCAR)
Brief Title: T Cells Expressing HER2-specific Chimeric Antigen Receptors(CAR) for Patients With HER2-Positive CNS Tumors
Acronym: iCAR
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Nabil Ahmed, Assistant Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-31973-iCAR
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Brain Tumor, Recurrent; Brain Tumor, Refractory
Keywords: CNS Tumors; T cells Expressing HER2-specific Chimeric Antigen Receptors; HER2-specific T cells; intracranial injection
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HER2-specific T cells - High Risk (Experimental): Subjects with HER2 staining of Grade 3 (51-100% of cells staining for HER2) and intensity scores of 3+ will be assigned to the High Risk arm. Three cell dosing schedules (1, 2, 3) consisting of combinations of three cell doses (A, B, C) will be evaluated.
  Interventions: Biological: HER2-specific T cells
- HER2-specific T cells - Standard Risk (Experimental): All other patients not meeting the high risk description will be assigned to the Standard Risk arm. Three cell dosing schedules (1, 2, 3) consisting of combinations of three cell doses (A, B, C) will be evaluated.
  Interventions: Biological: HER2-specific T cells

INTERVENTIONS:
Biological: HER2-specific T cells — Dosing Schedule 1:
  Cycle 1 A: 1x10^7 cells
  Cycle 2 A: 1x10^7 cells
  Cycle 3 A: 1x10^7 cells
  Dosing Schedule 2:
  Cycle 1 A: 1x10^7 cells
  Cycle 2 B: 3x10^7 cells
  Cycle 3 B: 3x10^7 cells
  Dosing Schedule 3:
  Cycle 1 A: 1x10^7 cells
  Cycle 2 B: 3x10^7 cells
  Cycle 3 C: 1x10^8 cells
  Subsequent cycles*
  *Additional cycles may be administered at ≤ the final cell dose reached in cycle 3, provided that the subject continues to meet eligibility criteria and does not have confirmed progressive disease.
  Other Names: Dosing Schedules 1, 2, and 3

SUMMARY:
This study is for patients that have brain cancer. The body has different ways of fighting infection and disease. No single way seems perfect for fighting cancers. This research study combines two different ways of fighting cancer: antibodies and T cells. Antibodies are types of proteins that protect the body from infectious diseases and possibly cancer. T cells, also called T lymphocytes, are special infection-fighting immune cells present in the blood that can kill other cells, including cells infected with viruses and tumor cells. Both antibodies and T cells have been used to treat patients with cancers. They have shown promise, but have not been strong enough to cure most patients.

The antibody used in this study is called anti-HER2 (Human Epidermal Growth Factor Receptor 2). This antibody sticks to tumor cells because of a substance on the outside of these cells called HER2. Many types of brain tumors are positive for HER2 . HER2 antibodies have been used to treat people with HER2-positive cancers. For this study, the HER2 antibody has been changed so that instead of floating free in the blood it is now attached to T cells. When an antibody is joined to a T cell in this way it is called a chimeric antigen receptor (CAR). These CAR-T cells seem to be able to kill tumors like the one these patients have, but they don't last very long and so their chances of fighting the cancer are limited. Therefore, developing ways to prolong the life of these T cells should help them fight cancer.

These HER2-CAR T cells are an investigational product not approved by the Food and Drug Administration.

The purpose of this study is to find the largest safe dose of HER2-CAR T cells, to learn what the side effects are, and to see whether this experimental intervention might help patients with brain tumors who volunteer to test this new agent.

DETAILED DESCRIPTION:
First, to find out if HER2 is expressed in the patient's brain cancer, the investigators will need to obtain the tissue block or tissue specimen that was used to make the original diagnosis. If there is enough material, investigators may also look for other proteins that may be targets for this sort of immune therapy in the future. Up to 90mls (18 tsp) of blood will be drawn on two occasions for a total of 180mls (36tsp). The total amount of blood drawn will not be more than 3 ml (less than 1 teaspoon) per 2.2 lbs of body weight.

To make HER2 CAR T cells the investigators will introduce the HER2 CAR gene into patient's T cells. To get the HER2 antibody to attach to the surface of the T cells, investigators will insert the antibody gene into the T cells. This is done with a virus called a retrovirus that has been made for this study and will carry the antibody gene into the T cell. This virus also helps the investigators find the T cells in patient's blood after they inject them. Most of the cells generated will be frozen and stored to give back to the patient.

This is a dose escalation study. This means that at the beginning, patients will be started on the lowest dosing schedule (1 of 3 different levels) of T cells. Once that dose schedule proves safe, the next group of patients will be started at a higher schedule. This process will continue until all 3 dose schedules are studied. If the side effects are too severe, the dose will be lowered or the T-cell infusions will be stopped.

The patient will be given three injections of cells two weeks apart into a special catheter that a neurosurgeon will implant into the tumor or the cavity left in the brain after surgical removal or into the fluid-filled space in your brain. The first injection of cells you receive will be the lowest dose. The subsequent injections, depending on the patient's assigned dosing schedule, may be higher than the first. Before the patient receives each injection, they may be given a dose of Tylenol. Each injection will take between 1 and 10 minutes. The patient will be admitted for overnight observation after each T-cell injection. Injections of T cells will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital or Houston Methodist Hospital.

If the patient has stable disease (the tumor did not grow), a reduction in the size of the tumor on imaging studies, or unconfirmed progressive disease, but health status is stable after the start of T-cell injections (at least 6 weeks after), they can receive additional doses of the T cells at 2 to 4 week intervals if they wish. Additional doses of T cells will be given at the highest cell dose the patient receives during the initial three cell infusions. Therefore, the dose the patient receives for additional doses may be higher than the initial dose they received.

Before being treated, the patient will receive a series of standard medical tests: physical exam, blood tests to measure blood cells, kidney and liver function,' pregnancy test if the patient is a female who could potentially become pregnant or might be pregnant, measurements of patient's tumor by routine imaging studies.

The patient will receive standard medical tests when they are getting the infusions and after: physical exams, blood tests to measure blood cells, kidney and liver function, measurements of patient's tumor by routine imaging studies 6 weeks after the infusion.

To learn more about the way the HER2-CAR T cells are working and how long they last in the body, an extra amount of blood, based on patient's weight, up to a maximum of 60 mL (12 teaspoons) of blood will be taken on the day of the T-cell infusion (before and 1 to 4 hours after the T-cell infusion), 3-4 days after the infusion (this one is optional), 1, 2, 4 and 6 weeks after the T-cell infusion and every 3 months for 1 year, every 6 months for 4 years, then yearly for a total of 15 years. This volume is considered safe, but may be decreased if the patient is anemic. This sample will be kept in a coded manner so that only the study staff may identify the patient.

During the time points listed above, if the T cells are found in patient's blood at a certain amount, an extra 5ml of blood may need to be collected for additional testing.

To see if there are any long-term side effects of gene transfer, the investigators will follow the patient up to 15 years.

If the patient receives additional T-cell infusions after the first one, s/he will have the same tests and blood draws as described above.

If the patient has a tumor biopsy or lumbar puncture to obtain CSF performed any time while s/he are on the study, a sample of this will be requested for research purposes.

If the patient develops a second abnormal growth, significant blood or nervous system disorder during the trial, a biopsy sample of the tissue will be tested for research purposes (if a sample can be obtained).

ELIGIBILITY:
Inclusion criteria at the time of procurement.

* Recurrent or refractory HER2 positive primary central nervous system (CNS) tumor or HER2 positive tumor metastatic to the CNS. Patients in whom tumor resection (gross total or subtotal resection) is medically feasible can undergo surgery after procurement and prior to treatment.
* Karnofsky/Lansky score of greater than or equal to 60
* Informed consent explained to, understood by and signed by subject/guardian. Subject/guardian given copy of informed consent

Exclusion Criteria at the time of procurement:

* Diagnosis of DIPG
* Bulky tumors causing midline shift and/or symptoms/signs due to impending herniation
* Known HIV positivity

Treatment Inclusion criteria:

* Recurrent or refractory HER2-positive* primary CNS tumor or HER2-positive solid tumor metastatic to the CNS

  * Immunohistochemistry (IHC) or RT-PCR will be used to determine HER2 positivity. Results will be compared to standard controls. HER2 expression in tumors on IHC should be greater than or equal to grade 1 and greater than or equal to 1+ intensity score. Wherein grades are defined as: Grade 0: no staining; Grade 1: 1-25%; Grade 2: 26-50% and Grade 3: 51-75% and Grade 4: 76-100% of cell staining for HER2 and intensity scores are: negative; 1+; 2+ and 3+ using breast cancer standard arrays as a guide for intensity.
* Intracranial catheter (such as Rickham or Ommaya) in place
* Age ≥ 3 years
* Life expectancy ≥ 6 weeks
* Karnofsky/Lansky score ≥ 60
* Bilirubin less than or equal to 3x upper limit of normal, AST less than or equal to 5x upper limit of normal, ALT less than or equal to 5x upper limit of normal, serum creatinine less than or equal to 2x upper limit of normal for age, and Hgb greater than or equal to 7.0 g/dL
* Pulse oximetry of greater than or equal to 90% on room air
* Sexually active subjects must be willing to utilize one of the more effective birth control methods for 6 months after the T cell infusion. The male partner should use a condom
* Available autologous transduced T lymphocytes with greater than or equal to 15% expression of HER2 CAR determined by flow-cytometry and killing of HER2-positive targets greater than or equal to 20% in cytotoxicity assay
* Patients who have undergone tumor resection should have recovered from the surgery. Patients with neurological deficits should have deficits that are stable for minimum of 1 week prior to treatment.
* Subjects should have been off other investigational antineoplastic therapy for two weeks prior to CAR T cell infusion. Temozolomide will be allowed up to 48 hours pre-infusion. Dexamethasone up to a total dose of 2 mg per day will be allowed if medically indicated
* Informed consent explained to, understood by and signed by research subjects/guardian. Subject/guardian given copy of informed consent.

Treatment Exclusion Criteria:

* Severe intercurrent infection
* Known HIV positivity
* Pregnant or lactating
* History of hypersensitivity reactions to murine protein-containing products.
* Diagnosis of DIPG
* Steroid dose of dexamethasone greater than 2 mg per day (or equivalent)

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2037-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicity after administration of autologous T cells expressing transgenic chimeric antigen receptors (CAR) targeting the HER2 molecule | 6 weeks
  To evaluate the safety of autologous T cells expressing transgenic chimeric antigen receptors (CAR) targeting the HER2 molecule administered into the tumor, tumor resection cavity, and/or cerebrospinal fluid (CSF) space of subjects with progressive recurrent or refractory HER2-positive primary central nervous system (CNS) tumor or HER2 positive tumor metastatic to the CNS, excluding diffuse intrapontine glioma (DIPG), after standard of care interventions.

SECONDARY OUTCOMES:
Number of Patients with a tumor response | 6 weeks
  To evaluate the effects of gene modified T cells on measurable disease.

CONTACTS AND LOCATIONS:
Overall Officials: Nabil M Ahmed, MD, Principal Investigator — Baylor College of Medicine - Texas Children's Hospital; Shoba Navai, MD, Principal Investigator — Baylor College of Medicine - Texas Children's Hospital; Meenakshi Hegde, MD, Principal Investigator — Baylor College of Medicine - Texas Children's Hospital
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas

DOCUMENTS (1):
  • Informed Consent Form (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT02442297/ICF_000.pdf